CLINICAL TRIAL: NCT04138017
Title: Clinical and Radiographic Outcomes Using ViviGen® Cellular Bone Matrix for Complex Hindfoot Arthrodesis
Brief Title: ViviGen Cellular Bone Matrix for Hindfoot or Ankle Arthrodesis
Acronym: ViviGen
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Joseph Park, Associate Professor, Department of Orthopaedic Surgery, University of Virginia
Other Study IDs: 20532
Record Dates: First submitted 2019-01-02; First posted 2019-10-24 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Ankle Deformity; Ankle Arthritis
Keywords: Arthrodesis
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ViviGen Cellular Bone Matrix: Patients will receive the vivigen cellular bone matrix
  Interventions: Device: ViviGen

INTERVENTIONS:
Device: ViviGen — A cellular bone matrix which includes viable osteoblasts within a corticocancellous and demineralized bone carrier, represents a unique alternative to autograft or existing products which utilize mesenchymal stem cells.

SUMMARY:
To evaluate the fusion status of the hindfoot bones after receiving the ViviGen graft, an FDA approved cellular bone matrix. This is used in a population indicated for hindfoot arthrodesis as an alternative to an autograft.

ELIGIBILITY:
Inclusion Criteria:

* Patient with prescribed standard of care unilateral hindfoot ankle arthrodesis procedure
* Age 18-80
* Willing to complete all follow up evaluations

Exclusion Criteria:

* Prior infection at site of planned arthrodesis
* Prior arthrodesis procedure
* Inability to maintain non-weight bearing status
* Bone defect requiring more than 10 cc of bone graft material
* Known Vitamin D deficiency with a Vitamin D level of <30ng/ml 1 week prior to surgery
* Inadequate bone stock to allow for rigid internal fixation
* Hemoglobin A1c greater than 8.0%
* Tobacco or Nicotine use 6 weeks prior to surgery
* BMI greater than 40

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in this study are receiving Vivigen as part of standard care. They are not assigned to receive Vivigen as part of study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Park, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ViviGen Cellular Bone Matrix
Started | 15
Completed | 14 (1 subject did not complete 2 of the time points and not included in final published data)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | ViviGen Cellular Bone Matrix
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.07 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Union Rates
Description: Radiographic evidence of successful arthrodesis confirmed on Computed Tomography (CT) scan defined by >50%. Results are for total number of joints fused which exceeds the number of participants due to some subjects having multiple joints fused.
Time Frame: 12 months
Population: total number of joints assessed for fusion.
Measure: Number; unit: joints fused
Units Other Than Participants: joints
Arm/Group | ViviGen Cellular Bone Matrix
Number analyzed (Participants) | 14
Number analyzed (joints) | 30
joints fused | 23

2. Secondary Outcome: Failure of Hardware or Obvious Non-union
Description: Failure measured through clinical and radiographic evidence
Time Frame: 12 months
Population: of the 30 joints analyzed in 14 subjects, 7 did not fuse to 50%
Measure: Number; unit: participants
Units Other Than Participants: joints
Arm/Group | ViviGen Cellular Bone Matrix
Number analyzed (Participants) | 14
Number analyzed (joints) | 30
participants | 7

3. Secondary Outcome: Foot and Ankle Ability Measure (FAAM) - Activities of Daily Living (ADL) Subscale
Description: For this study, the researchers only utilized the ADL subscale. This patient-reported outcome measure is a 21-item questionnaire assessing fundamental mobility and daily activities. Responses use a 5-point Likert scale ranging from 4 (no difficulty) to 0 (unable to do), with N/A responses excluded. The responses are summed, and the total possible score is calculated by multiplying the number of answered items by 4 (maximum score: 84). The total score is divided by the highest potential score, then multiplied by 100 to yield a percentage. Higher percentages indicate greater physical function, with 100% representing no functional limitations, on the ADL subscale.
Time Frame: baseline, 3 month, 6 month, 1 year
Population: 1 subject did not complete the 1 year time point.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | ViviGen Cellular Bone Matrix
Number analyzed (Participants) | 14
Percentage
  baseline | 53.52 (18.94)
  3 month | 61.09 (23.76)
  6 month | 73.30 (20.86)
  1 year: number analyzed (Participants) | 13
  1 year | 80.69 (18.69)

4. Secondary Outcome: Vitamin D Levels
Description: 25-Hydroxyvitamin D is the primary circulating form of vitamin D and is the most commonly used measure to assess vitamin D status in the blood. The reference range for 25-hydroxy vitamin D test is 20-80 ng/mL. A low test level would indicate lower concentrations of Vitamin D.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ViviGen Cellular Bone Matrix
Number analyzed (Participants) | 14
ng/mL
  Baseline | 48.17 (14.99)
  6 month | 55.86 (15.00)

5. Secondary Outcome: American Orthopaedic Foot and Ankle Society(AOFAS) Hindfoot Score
Description: Patient reported outcome for a standardized evaluation of clinical status of ankle- hindfoot. Patient reports their pain and the physician records physical assessment of alignment. Finally function is reported and the AOFAS score ranged from 0-100 with 100 being healthy ankles.
Time Frame: baseline, 3 month, 6 month, 1 year
Population: 1 subject did not complete 1 year timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ViviGen Cellular Bone Matrix
Number analyzed (Participants) | 14
score on a scale
  baseline | 48.93 (12.93)
  3 month | 64.71 (13.38)
  6 month | 69.43 (21.86)
  1 year: number analyzed (Participants) | 13
  1 year | 79.85 (12.23)

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | ViviGen Cellular Bone Matrix
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ViviGen Cellular Bone Matrix (N=15)
Revision surgery of Triple Arthrodesis, hardware removal (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ViviGen Cellular Bone Matrix (N=15)
Left ankle synovitis / impingement (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04138017/Prot_SAP_000.pdf